CLINICAL TRIAL: NCT00521651
Title: Physical Activity and Its Components in Relation to Plasma Inflammatory Markers of Cancer Risk Among Chinese Adults
Brief Title: PRelationship Between Physical Activity and Cancer Ris
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905190; 05-C-N190; NCT00340067 (obsolete NCT alias)
Record Dates: First submitted 2007-08-25; First posted 2007-08-28 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Cancer
Keywords: Physical Activity; Cancer Risk
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Community Cohort: Men and Women from two Shanghai cohort studies.

SUMMARY:
This protocol is a sub-study of the ongoing "Protect Health and Reduce Cancer Risk" study conducted in Shanghai, China, and sponsored by the Shanghai Cancer Institute, Vanderbilt University, and the National Cancer Institute. The parent study is designed to examine the relationship of diet, lifestyle, occupational, and environmental risk factors, as well as genetic variation, to cancer incidence in a large cohort of men in women between 40 and 70 years of age. The current sub-study will assess the validity and reliability of a new physical activity questionnaire for use in the parent study and to evaluate whether different types of activity and the frequency, intensity, and duration of activity are associated with markers that have been linked to cancer risk, such as C-reactive protein, interleukin 6 and soluble tumor necrosis factor alpha.

Participants in the current 12-month study are selected from among men and women participating in the "Protect Health and Reduce Cancer Risk" study. Participants keep a diary of their physical activity and complete two 30-minute interviews about their physical activity, one at the beginning and one at the end of the study period. Every 3 months for 7 consecutive days, they wear a pager-sized activity monitor on their waist that records their physical activity patterns during that period of time. They provide blood and urine samples four times during the study and, at the end of the study, undergo a health examination that includes an electrocardiogram, body composition measurement, and physical fitness test. The fitness test is a step-test consisting of 3-minute stages in which the subject successively increases the stepping speed until reaching 85 percent of his or her predicted maximal heart rate.

Blood and urine samples are analyzed for levels of nutrients and certain proteins, and are stored for future studies related to nutrition and physical activity and possibly for genetic studies related to health, nutrition, exercise, or disease.

DETAILED DESCRIPTION:
In the past decade, China has experienced fundamental decreases in the populations' physical activity levels, due to increasingly sedentary occupations and lifestyles. However, the transition to a Western lifestyle has not reached the entire Chinese population. The resulting wide range of between-person variation in physical activity provides an unparalleled opportunity for physical activity studies. Although physical activity measurement techniques have evolved considerably over the past years, the main obstacle in quantifying physical activity is the complexity of precisely measuring its individual components, particularly low to moderate-intensity activities.

Recently, investigators at Vanderbilt University, the Shanghai Cancer Institute, and the DCEG initiated two prospective population-based cohort studies: the Shanghai Women's Cohort and the Shanghai Men's Cohort. The aim of these studies is to prospectively examine the relations of diet, lifestyle, occupational, and environmental risk factors, as well as genetic variation, to cancer incidence among 75,000 women and 73,000 men, aged 40 to 70 years old, and residing in Shanghai, China. We propose to conduct a study among 600 women and men participating in these two cohort studies. The specific objectives of the current study are to develop a comprehensive physical activity questionnaire and to assess the validity and reliability of this instrument in the Shanghai cohorts using objective measures of physical activity/physical fitness: activity monitors, and the Modified Canadian Aerobic Fitness Test. In addition, we intend to evaluate whether different types and parameters of physical activity are associated with circulating levels of specific inflammatory markers that have been linked to cancer risk. The specific markers are C-reactive protein (CRP), interleukin 6 (IL-6), and soluble tumor necrosis factor alpha (TNF-a). The impact of potentially confounding variables of the association between physical activity and inflammatory markers, such as recent exercise, use of anti-inflammatory drugs, and current or recent infections, will be carefully accounted for in the analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:

The current study will be conducted in random sub samples of the Shanghai Women's Cohort Study and Shanghai Men's Cohort Study. Eligibility in these 2 cohort studies was determined based on the following: 40 to 70 years of age and residing in one of 7 Shanghai urban areas that is representative of all of urban Shanghai. Both women and men will be included in the study. No exclusions will be made by race, although it should be noted that the study population of the Shanghai Women's Cohort and Shanghai Men's Cohort Study is virtually 100% Asian.

EXCLUSION CRITERIA:

There wil be no prior from participation, other than the presence of physical ailments preventing subjects from participating in the study. Before participating in the fitness test, subjects will be screened for cardiovascular disease, othopedic limitations, or other factors that contraindicate testing, including pregnancy, respiratory problems at rest (labored breathing or persistent cough), presence of illness or fever, or swelling of the lower extremities. In addition, participants who do not adhere to the pre-test instructions of not eating heavily or drinking alcohol 2 hours before the test will be excluded from performing the fitness test.

Children will not be included in the current study, because study subjects are comprised of participants in the Shanghai Womens's Cohort Study and the Shanghai Men's Cohort Study, who are 40 to 70 years of age.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2005-08-01 (Actual); Primary Completion 2009-04-23 (Actual); Study Completion 2009-04-23 (Actual)

PRIMARY OUTCOMES:
Physical activity behaviors and circulating or excreted biomarkers | 1 Year
  Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Matthews, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- Vanderbilt University, Nashville, Tennessee, United States
- Shanghai National Cancer Institute, Shanghai, China

REFERENCES:
- [Background] McTiernan A, Ulrich C, Slate S, Potter J. Physical activity and cancer etiology: associations and mechanisms. Cancer Causes Control. 1998 Oct;9(5):487-509. doi: 10.1023/a:1008853601471. PMID 9934715
- [Background] Friedenreich CM. Physical activity and cancer prevention: from observational to intervention research. Cancer Epidemiol Biomarkers Prev. 2001 Apr;10(4):287-301. PMID 11319168
- [Background] Popkin BM. The nutrition transition and obesity in the developing world. J Nutr. 2001 Mar;131(3):871S-873S. doi: 10.1093/jn/131.3.871S. PMID 11238777